CLINICAL TRIAL: NCT00835003
Title: Timing of Elective Caesarean Section and Neonatal Morbidity - a Randomised Multicentre Study
Brief Title: Timing of Planned Caesarean Section and Morbidity of the Newborn
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Julie Glavind, MD, PhD, Aarhus University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: AAUH091077
Record Dates: First submitted 2009-02-02; First posted 2009-02-03 (Estimated); Results first posted 2014-07-03 (Estimated); Last update posted 2014-07-03 (Estimated); Status verified 2014-06

CONDITIONS: Respiratory Disorders; Intensive Care, Neonatal
Keywords: Neonatal admission; Elective Caesarean Section; Timing; Choice behavior; Intraoperative complications; Postoperative complications
MeSH Terms: conditions — Respiration Disorders; Intraoperative Complications; Postoperative Complications | interventions — Elective Surgical Procedures

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Elective caesarean section at 38 weeks and 3 days of gestation
  Interventions: Procedure: Elective caesarean section
- 2 (Active Comparator): Elective caesarean section at 39 weeks and 3 days of gestation
  Interventions: Procedure: Elective caesarean section

INTERVENTIONS:
Procedure: Elective caesarean section — Procedure performed at 38 weeks and 3 days of gestation (+/- 2 days)
  Other Names: Elective surgery; Planned caesarean section
  Arms: 1
Procedure: Elective caesarean section — Procedure performed at 39 weeks and 3 days of gestation (+/- 2 days)
  Other Names: Elective surgery; Planned caesarean section
  Arms: 2

SUMMARY:
The caesarean section rate is rising globally. About 10% of the newborns are submitted to a neonatal department after planned caesarean section, primarily with respiratory disorders. More children are submitted if caesarean is performed earlier in pregnancy.

Study hypothesis: More newborns are admitted after planned caesarean at 38 weeks and 3 days of gestation than after 39 weeks and 3 days of gestation.

Aim of study: To compare elective caesarean section performed at 38 weeks and 3 days of gestation with 39 weeks and 3 days of gestation. According to this timing to determine the proportion of newborns admitted within 48 hours after birth.

ELIGIBILITY:
Inclusion Criteria:

* Elective caesarean section
* Gestational age determined at 12 weeks ultrasound scan
* Singleton pregnancy

Exclusion Criteria:

* < 18 years of age (at time of randomization)
* In need of an interpreter to communicate in danish
* Diabetes, both gestational and before pregnancy
* A mother with an estimated high risk of caesarean section before 39+5 weeks

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1273 (Actual)
Dates: Start 2009-03; Primary Completion 2011-11 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julie Glavind, MD, Principal Investigator — Department of Gynecology and Obstetrics, Aarhus University Hospital Skejby; Niels Uldbjerg, MD,Professor, Study Chair — Department og Gynecology and Obstetrics, Aarhus University Hospital Skejby; Tine B Henriksen, MD, Professor, Study Chair — Neonatal Department, Aarhus University Hospital Skejby; Sara F Kindberg, PhD, midwife, Study Chair — Perinatal Research Unit, Aarhus University Hospital Skejby
Locations (7):
- Denmark (7):
  - University Hospital of Odense, Odense, Odense
  - Aarhus University Hospital, Aalborg Hospital, Aalborg
  - Department of Obstetrics and Gynecology, Aarhus University Hospital Skejby, Aarhus N
  - Regional Hospital of Herning, Herning
  - Hospital of Kolding, Kolding
  - Regional Hospital of Randers, Randers
  - Regional Hospital of Viborg, Viborg

REFERENCES:
- [Derived] Glavind J, Henriksen TB, Kindberg SF, Uldbjerg N. Randomised trial of planned caesarean section prior to versus after 39 weeks: unscheduled deliveries and facility logistics--a secondary analysis. PLoS One. 2013 Dec 20;8(12):e84744. doi: 10.1371/journal.pone.0084744. eCollection 2013. PMID 24376842
- [Derived] Glavind J, Kindberg SF, Uldbjerg N, Khalil M, Moller AM, Mortensen BB, Rasmussen OB, Christensen JT, Jorgensen JS, Henriksen TB. Elective caesarean section at 38 weeks versus 39 weeks: neonatal and maternal outcomes in a randomised controlled trial. BJOG. 2013 Aug;120(9):1123-32. doi: 10.1111/1471-0528.12278. Epub 2013 May 20. PMID 23682628

RESULTS

PARTICIPANT FLOW:
Groups:
- 38 Weeks Group: Elective caesarean section at 38 weeks and 3 days of gestation
  Elective caesarean section: Procedure performed at 38 weeks and 3 days of gestation (+/- 2 days)
- 39 Weeks Group: Elective caesarean section at 39 weeks and 3 days of gestation
  Elective caesarean section: Procedure performed at 39 weeks and 3 days of gestation (+/- 2 days)
Period: Overall Study
Arm/Group | 38 Weeks Group | 39 Weeks Group
Started | 636 | 638
Completed | 636 | 638
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 38 Weeks Group | 39 Weeks Group | Total
Number analyzed (Participants) | 636 | 638 | 1274
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.1 (4.4) | 31.6 (4.6) | 31.8 (4.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 636 | 638 | 1274
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Denmark | 636 | 638 | 1274

OUTCOME MEASURES:

1. Primary Outcome: Neonatal Admission After Elective Caesarean Section
Time Frame: 48 hours
Measure: Number; unit: participants
Arm/Group | 38 Weeks Group | 39 Weeks Group
Number analyzed (Participants) | 635 | 637
participants | 88 | 76
Statistical Analysis 1: Comparison: 38 Weeks Group vs 39 Weeks Group; Test type: Non-Inferiority or Equivalence — Power calculations estimated a sample size of 1272 women with an estimated proportion of 8% in the 39 weeks Group and 14% in the 38 weeks group; p = 0.31, Chi-squared; Risk Ratio (RR) = 0.86, 95% CI 2-sided [0.65 to 1.15]

2. Secondary Outcome: Neonatal Diagnoses
Time Frame: 30 days
Reporting Status: Not Posted

3. Secondary Outcome: Duration of Neonatal Treatment With Ventilator, CPAP, Oxygen and/or Antibiotics
Time Frame: 30 days
Reporting Status: Not Posted

4. Secondary Outcome: Maternal Haemorrhage in ml or Organ Laceration During Caesarean Section.
Time Frame: 30 days
Reporting Status: Not Posted

5. Secondary Outcome: Maternal Fever, Wound Infection, Need of Wound Operative Revision and Antibiotics, Duration of Admission
Time Frame: 30 days
Reporting Status: Not Posted

6. Secondary Outcome: Maternal Satisfaction With Timing of Elective Caesarean Section
Time Frame: 2 months
Reporting Status: Not Posted

7. Secondary Outcome: Post Partum Depression
Time Frame: 2 months
Reporting Status: Not Posted

8. Secondary Outcome: Pediatric Admission and Morbidity
Time Frame: 2 months post partum
Reporting Status: Not Posted

9. Secondary Outcome: Pediatric Admission and Morbidity
Time Frame: From birth until 2 years of age
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | 38 Weeks Group | 39 Weeks Group
Serious Adverse Events (participants affected / at risk) | 1/636 | 2/638
Other Adverse Events (participants affected / at risk) | 0/636 | 0/638
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 38 Weeks Group (N=636) | 39 Weeks Group (N=638)
Fetal death (Pregnancy, puerperium and perinatal conditions) | 1 | 1
Neonatal death (Respiratory, thoracic and mediastinal disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes